CLINICAL TRIAL: NCT03464084
Title: Interaction of Melatonin and Light With MTNR1B Genotype on Glucose Control - Study 2
Brief Title: Interaction of Melatonin With MTNR1B Genotype on Glucose Control - Study 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Frank AJL Scheer, PhD, Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2015P000857B; R01DK102696 (NIH)
Record Dates: First submitted 2018-03-02; First posted 2018-03-13 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Glucose; Circadian Rhythm; Melatonin; Genes; Light
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- bright light placebo (Other)
  Interventions: Drug: placebo; Other: bright light
- bright light melatonin (Other)
  Interventions: Dietary Supplement: melatonin; Other: bright light
- dim light (Other)
  Interventions: Other: dim light

INTERVENTIONS:
Drug: placebo — Capsules containing microcrystalline cellulose
  Arms: bright light placebo
Dietary Supplement: melatonin — 5 mg of melatonin per os.
  Arms: bright light melatonin
Other: bright light — room light will be bright
  Arms: bright light melatonin; bright light placebo
Other: dim light — room light will be dim
  Arms: dim light

SUMMARY:
This project aims to test the impact of melatonin and MTNR1B variation on regulation glucose regulation in a highly controlled in-laboratory setting and ex vivo in pancreatic islets.

DETAILED DESCRIPTION:
The investigators' recent GWAS discovery of MTNR1B as a novel type 2 diabetes gene has sparked great interest into the role of melatonin in glycemic control, for which the mechanism is largely unknown. This research will determine the effect of melatonin and MTNR1B on glycemic control under highly-controlled, in-laboratory protocols while manipulating circulating melatonin concentrations (both up and down) and assessing glycemic control by frequently-sampled intravenous glucose tolerance tests, as well as in ex vivo human pancreatic islets. This research will provide mechanistic insights into the metabolic effects of melatonin and the MTNR1B risk variant and may help in evidence-based approaches and personalized recommendations to improve glycemic control in night shift workers and late-night eaters.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index: 20 and 35 kg/m2
* Age: 21-55 years of age
* Caucasian
* Non-smoking
* With regular sleep-wake cycle
* Passed medical and psychological screening tests

Exclusion Criteria:

* Acute, chronic or debilitating medical conditions
* History of neurological or psychiatric disorder
* History of sleep disorder or regular use of sleep-promoting medication
* Current prescription, herbal, or over-the-counter medication use
* Traveling across 2 or more time zones within past 3 months
* Worked night or rotating shift work within past 1 year
* Drug or alcohol dependency

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-02-17 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2022-07-19 (Actual)

PRIMARY OUTCOMES:
change in glucose tolerance | Day 1 of the three in-lab protocols
  glucose responses to test meal compared across the three in-lab protocols

SECONDARY OUTCOMES:
change in first-phase insulin release | Day 1 of the three in-lab protocols
  insulin responses to test meal compared across the three in-lab protocols

CONTACTS AND LOCATIONS:
Overall Officials: Frank AJL Scheer, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States